CLINICAL TRIAL: NCT00833092
Title: Magnesium Nutrition and Sleep Behavior in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GFHNRC014
Record Dates: First submitted 2009-01-27; First posted 2009-01-30 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Nutritional Deficiency; Insomnia
Keywords: magnesium; Nutritional Requirements; Sleep
MeSH Terms: conditions — Malnutrition; Sleep Initiation and Maintenance Disorders | interventions — Sugars; Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator): Sugar Pill
  Interventions: Dietary Supplement: Sugar Pill
- magnesium (Active Comparator): 300 milligrams of magnesium daily
  Interventions: Dietary Supplement: magnesium

INTERVENTIONS:
Dietary Supplement: Sugar Pill — Sugar pill supplementation for 9 weeks
  Arms: Sugar pill
Dietary Supplement: magnesium — 300 milligrams daily for 8 weeks
  Arms: magnesium

SUMMARY:
Insomnia is not a natural part of aging but is higher in older adults because of a variety of factors common in later life. One of these factors may be a deficient magnesium status. This study will look at whether or not magnesium supplementation will improve sleep.

DETAILED DESCRIPTION:
Insomnia affects approximately one-third of older Americans. More than half of all people aged 65 and older experience sleep problems. The prevalence of insomnia and other sleep disorders is not a natural part of aging but is high in older adults because of a variety of factors common in late life. One of those factors may be a deficient magnesium status. There is a close association between sleep architecture, especially slow wave sleep, and activity in the glutamatergic and gamma-aminobutyric acid (GABA) system. Because magnesium is a natural N-methyl-D-aspartate (NMDA)antagonist and GABA agonist, magnesium apparently plays a key role in the regulation of sleep. Such a role is supported by supplementation, correlation, and animal studies showing that magnesium intake or status affects sleep organization.

ELIGIBILITY:
Inclusion Criteria:

* have sleep complaints
* Score greater than 5 on Pittsburgh Global Sleep Quality Index

Exclusion Criteria:

* taking medications that affect sleep
* taking 100 milligrams or more of magnesium
* body mass index of 40 or higher
* abnormal breathing conditions

Min Age: 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Forrest H Nielsen, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Background] Foley DJ, Monjan AA, Brown SL, Simonsick EM, Wallace RB, Blazer DG. Sleep complaints among elderly persons: an epidemiologic study of three communities. Sleep. 1995 Jul;18(6):425-32. doi: 10.1093/sleep/18.6.425. PMID 7481413
- [Background] Hunt CD, Johnson LK. Magnesium requirements: new estimations for men and women by cross-sectional statistical analyses of metabolic magnesium balance data. Am J Clin Nutr. 2006 Oct;84(4):843-52. doi: 10.1093/ajcn/84.4.843. PMID 17023712
- [Background] Ford ES, Mokdad AH. Dietary magnesium intake in a national sample of US adults. J Nutr. 2003 Sep;133(9):2879-82. doi: 10.1093/jn/133.9.2879. PMID 12949381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 2007 and 2008 by the USDA Grand Forks Human Nutrition Research Center staff in North Dakota.
Pre-assignment Details: 425 applications were received. 215 people did not meet the eligibility criteria. 99 people withdrew their application. 111 people were assigned to groups.
Groups:
- Sugar Pill: zero magnesium supplementation
Period: Overall Study
Arm/Group | Sugar Pill | Magnesium
Started | 54 | 57
Completed | 50 | 50
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Diarrhea | 0 | 2
Not completed — constipation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Magnesium | Total
Number analyzed (Participants) | 54 | 57 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 49 | 89
  >=65 years | 14 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.7) | 58.2 (6.2) | 59.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 43 | 82
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 54 | 57 | 111

OUTCOME MEASURES:

1. Primary Outcome: Global Pittsburgh Sleep Quality Index
Description: Improvement in the Pittsburgh Global Sleep Quality Index (PGQI). The index is based on a score of 0 to 21, the lower the score on the index the better the subject perceives their sleep.
Time Frame: 9 weeks
Population: Data from 4 participants (3 on sugar pill, 1 on magnesium) were omitted from statistical analysis because of protocol violations discovered near end of study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sugar Pill | Magnesium
Number analyzed (Participants) | 47 | 49
score on a scale | 6.30 (0.37) | 6.96 (0.36)

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Magnesium
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/57
Other Adverse Events (participants affected / at risk) | 0/54 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No